CLINICAL TRIAL: NCT00908882
Title: Telehealth Care Management and Tobacco Cessation for Veterans With PTSD
Brief Title: Tobacco Cessation for Veterans With Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NRI 08-117; COMIRB 08-0556 (Other: University of Colorado)
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Tobacco Use Cessation; Post Traumatic Stress Disorders
Keywords: Nursing Care; Veterans
MeSH Terms: conditions — Tobacco Use Cessation; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced PTSD Health Buddy and Motivational Interviewing (Experimental): Veterans with PTSD who smoke are exposed to an intervention which included a 90-day smoking cessation curriculum that is integrated into the PTSD Health Buddy Program and weekly motivational interviewing counseling by a nurse plus usual smoking cessation care
  Interventions: Behavioral: Motivation Interviewing Counseling
- Usual PTSD Health Buddy Care (No Intervention): Veteran with PTSD who smoke randomly assigned to this arm received standard of care for smoking cessation and used the standard PTSD Health Buddy

INTERVENTIONS:
Behavioral: Motivation Interviewing Counseling — Stage-based smoking cessation information written in the spirit of motivational interviewing in addition to weekly telephonic motivational interviewing counseling sessions
  Arms: Enhanced PTSD Health Buddy and Motivational Interviewing

SUMMARY:
The goal of this study is to improve the effectiveness of tobacco cessation treatment for veterans with Post Traumatic Stress Disorder (PTSD) through ongoing, integrated care management approach using telehealth and motivational interviewing counseling. Both tobacco dependence and PTSD represent enormous challenges to the Veterans Affairs (VA) healthcare system.

DETAILED DESCRIPTION:
Background: Veterans smoke at a higher rate (30%) than the U.S. adult population (21%), and veterans with PTSD have even higher rates of smoking (53-66%). Evidence has shown that any tobacco dependence treatment strategy must be integrated in the health care system because consistent and effective delivery of tobacco cessation requires coordinated interventions. Persistent tobacco users typically cycle through multiple periods of relapse and remission. Veterans with PTSD (279,256 in 2005) who are treated for smoking cessation may need more comprehensive aid to be successful. Failure to appreciate the chronic nature of tobacco dependence may impede comprehensive and consistent treatment. Care management using telehealth has been shown to improve access to care while reducing costs for veterans with chronic diseases and has the potential to coordinate smoking cessation with care for other chronic diseases. Nurses have successfully managed chronic diseases using telehealth by focusing on increasing self-management, positive behaviors and knowledge. Nurses are vital to increasing the level of support in the community through education and motivation and by responding to medical events in order to improve veterans' health.

Objectives: The study is designed to determine if adding motivational counseling and care management using the PTSD Health Buddy to usual care improves smoking quit rates of veterans with PTSD. Specific Aims are to compare: 1) self-reported quit attempts, progression through the stages of change, and quit rates, 2) patient perception of care coordination, and 3) changes in PTSD symptoms in veteran smokers with PTSD who receive a nurse-driven telephonic motivational counseling intervention triggered by responses to stage-based smoking cessation questions in addition to usual care to those who receive usual care only.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders IV criteria (DSM-IV) for diagnosis code 309.81 PTSD
* Willingness to participate
* Currently smoking 1 or more cigarettes per day

Exclusion Criteria:

* Use smokeless tobacco, pipes or cigars instead of cigarettes
* Have imminent risk of suicide or violence
* Have severe psychiatric symptoms or psychosocial instability likely to prevent participation in protocol (provider will assess appropriateness)
* Have clinically apparent gross cognitive impairment
* Unable to connect Health Buddy in home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2009-07; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Battaglia, PhD MS BS, Principal Investigator — Denver VA Medical Center
Locations (1):
- VA Eastern Colorado Health Care System, Denver, Denver, Colorado, United States

REFERENCES:
- [Result] Battaglia C, Stein KF. A clinical translation of the research article titled "Building a tobacco cessation telehealth care management program for veterans with posttraumatic stress disorder". J Am Psychiatr Nurses Assoc. 2013 Mar-Apr;19(2):92-7. doi: 10.1177/1078390313485907. No abstract available. PMID 23644676
- [Result] Battaglia C, Benson SL, Cook PF, Prochazka A. Building a tobacco cessation telehealth care management program for veterans with posttraumatic stress disorder. J Am Psychiatr Nurses Assoc. 2013 Mar-Apr;19(2):78-91. doi: 10.1177/1078390313483314. PMID 23644675
- [Derived] Peterson J, Prochazka AV, Battaglia C. Smoking cessation and care management for veterans with posttraumatic stress disorder: a study protocol for a randomized controlled trial. BMC Health Serv Res. 2015 Feb 1;15:46. doi: 10.1186/s12913-015-0706-6. PMID 25638351

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced PTSD Health Buddy and Motivational Interviewing: Veterans with PTSD who smoke and are exposed to a 90-day smoking cessation curriculum that is integrated into the PTSD Health Buddy Program and weekly motivational interviewing counseling by a nurse plus usual smoking cessation care
  Motivation Interviewing Counseling: Stage-based smoking cessation information written in the spirit of motivational interviewing in addition to weekly telephonic motivational interviewing counseling sessions
- Usual PTSD Health Buddy Care: Veteran with PTSD who smoke and receive standard of care for smoking cessation and use the standard PTSD Health Buddy
Period: Overall Study
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Started | 89 | 89
Completed | 61 | 59
Not Completed | 28 | 30

BASELINE CHARACTERISTICS:
Population: Arm 2 - 3 participants were found to be ineligible after signing consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care | Total
Number analyzed (Participants) | 89 | 86 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11.2) | 57 (10.8) | 55.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 74 | 77 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 77 | 77 | 154
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 72 | 72 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 89 | 86 | 175
Post Traumatic Stress Disorder Checklist [Mean (Standard Deviation); unit: units on a scale] — Range 17-85; > 50 indicates PTSD diagnosis
  units on a scale | 57 (11.9) | 60 (11) | 58.8 (11.5)
Geriatric Depression Scale [Mean (Standard Deviation); unit: units on a scale] — Range 1-15; > 6 indicates probably depression
  units on a scale | 8.9 (3.7) | 9.2 (3.8) | 9.1 (3.7)
Fagerstrom Test of Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — 0-3 low dependence 4-6 medium dependence 7-10 high dependence
  units on a scale | 5.4 (2) | 5 (2.3) | 5.3 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Quit Attempts - The Primary Outcome is the Number of Veteran's Who Make a Self-reported Quit Attempt (as Defined as a 24-hour Point Prevalence Rate).
Time Frame: During 90-session intervention period
Measure: Number; unit: participants
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 89 | 86
participants | 34 | 28

2. Primary Outcome: Number of Participants Who Progressed Along the Stage of Change Toward Action as Measured by the Transtheoretical Model of Change (Short Form) Questionnaire. This Will Identify Current Stage of Change for Each Subject.
Description: Transtheoretical Model of Change questionnaire:
  Are you currently a smoker?
  * Yes, I currently smoke (move to For Smokers Only section)
  * No, I quit within the last 6 months (ACTION STAGE)
  * No, I quit more than 6 months ago (MAINTENANCE STAGE)
  * No, I have never smoked (NONSMOKER) (For smokers only) In the last year, how many times have you quit smoking for at least 24 hours?
  (For smokers only) Are you seriously thinking of quitting smoking?
  * Yes, within the next 30 days (PREPARATION STAGE if they have one 24-hour quit attempt in the past year - refer to previous question... if no quit attempt then CONTEMPLATION STAGE)
  * Yes, within the next 6 months (CONTEMPLATION STAGE)
  * No, not thinking of quitting (PRECONTEMPLATION STAGE)
Time Frame: During 90-session intervention period
Measure: Number; unit: participants
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 89 | 86
participants | 36 | 35

3. Primary Outcome: Seven-day Point Prevalence -A Primary Outcome is the Number of Veteran's Who Self-reported Quit Smoking for Seven Days.
Time Frame: During 90-session intervention period
Measure: Number; unit: participants
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 89 | 86
participants | 20 | 22

4. Primary Outcome: Self-reported Quit Attempts - The Primary Outcome is the Number of Veteran's Who Make a Self-reported Quit Attempt (as Defined as a 24-hour Point Prevalence Rate).
Time Frame: During the 6-month follow-up period
Measure: Number; unit: participants
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 89 | 86
participants | 24 | 31

5. Primary Outcome: Seven-day Point Prevalence -A Primary Outcome is the Number of Veteran's Who Self-reported Quit Smoking for Seven Days.
Time Frame: During the 6-month follow-up period
Measure: Number; unit: participants
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 89 | 86
participants | 21 | 20

6. Primary Outcome: Number of Participants Who Progressed Along the Stage of Change Toward Action as Measured by the Transtheoretical Model of Change (Short Form) Questionnaire. This Will Identify Current Stage of Change for Each Subject.
Description: Are you currently a smoker?
  * Yes, I currently smoke (move to For Smokers Only section)
  * No, I quit within the last 6 months (ACTION STAGE)
  * No, I quit more than 6 months ago (MAINTENANCE STAGE)
  * No, I have never smoked (NONSMOKER) (For smokers only) In the last year, how many times have you quit smoking for at least 24 hours?
  (For smokers only) Are you seriously thinking of quitting smoking?
  * Yes, within the next 30 days (PREPARATION STAGE if they have one 24-hour quit attempt in the past year - refer to previous question... if no quit attempt then CONTEMPLATION STAGE)
  * Yes, within the next 6 months (CONTEMPLATION STAGE)
  * No, not thinking of quitting (PRECONTEMPLATION STAGE)
Time Frame: During the 6-month follow-up period
Measure: Number; unit: participants
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 89 | 86
participants | 22 | 21

7. Secondary Outcome: Post Traumatic Stress Disorder Checklist
Description: range 17-85; >50 indicates PTSD diagnosis
Time Frame: At end of 90-session intervention period
Population: These numbers represent those that completed the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 62 | 59
units on a scale | 54.5 (13.2) | 55.9 (13.5)

8. Secondary Outcome: Post Traumatic Stress Disorder Checklist
Description: range 17-85; >50 indicates PTSD diagnosis
Time Frame: At the end of the 6-month follow-up period
Population: These numbers represent those that completed the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 61 | 59
units on a scale | 58.4 (11.4) | 62.4 (10.9)

9. Secondary Outcome: Geriatric Depression Scale
Description: range 1-15; >6 indicates depression
Time Frame: At the end of the 90-session intervention period
Population: These numbers represent those that completed the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 68 | 62
units on a scale | 7.9 (4.2) | 10 (4.2)

10. Secondary Outcome: Geriatric Depression Scale
Description: range 1-15; >6 indicates depression
Time Frame: At the end of the 6-month follow-up period
Population: These numbers represent those who completed the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Number analyzed (Participants) | 61 | 59
units on a scale | 8.4 (4.2) | 9.8 (3.8)

ADVERSE EVENTS:
Groups:
- Usual PTSD Health Buddy Care: Veteran with PTSD who smoke received standard of care for smoking cessation and use the standard PTSD Health Buddy
Arm/Group | Enhanced PTSD Health Buddy and Motivational Interviewing | Usual PTSD Health Buddy Care
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 0/89 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes